CLINICAL TRIAL: NCT01522677
Title: A Phase I/II Study of Neoadjuvant Photodynamic Immunomodulation for Colon Cancer
Brief Title: A Study of Neoadjuvant Photodynamic Immunomodulation for Colon Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Edward Nelson (Other)
Collaborators: University of California, Irvine (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Edward Nelson, Dr. Edward Nelson, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 10-26; 1R21CA153594 (NIH)
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Colon Cancer
Keywords: tumor immunology; neoadjuvant; colonoscopy; photosensitization
MeSH Terms: conditions — Colonic Neoplasms; Photosensitivity Disorders | interventions — 1-phenyl-3,3-dimethyltriazene; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PDT (Experimental): Participants receive neoadjuvant 5-ALA and PDT.
  Interventions: Drug: PDT with 5-ALA radiosensitization

INTERVENTIONS:
Drug: PDT with 5-ALA radiosensitization — Patients receive neoadjuvant PDT with radiosensitizing 5-ALA 4 days prior to surgery for colon cancer.
  Other Names: Photodynamic therapy; 5-ALA

SUMMARY:
The central hypothesis for this study is that it is safe and feasible to administer intraluminal photodynamic therapy (PDT) to colon cancers by colonoscopy to induce localized inflammatory/immune response. The objective is to demonstrate the feasibility and safety of PDT to colon cancer patients administered before surgery and to characterize the inflammatory/immune response at the tumor site and systemically. The long-term objective of these studies is to modify he natural biology of colorectal cancers and improve patient survival.

DETAILED DESCRIPTION:
The central hypothesis for this study is that it is safe and feasible to administer intraluminal photodynamic therapy (PDT) to colon cancers, via colonoscopy, in the neoadjuvant setting to induce localized tumor cell death and an inflammatory/immune response with an increased Th1 component, utilizing 5-ALA as a photosensitizer. The objective is to conduct an initial phase I/II clinical study to demonstrate the feasibility and safety of colonoscopic, neoadjuvant intraluminal PDT to colon cancer patients administered 96 hours pre-resection, to characterize the inflammatory/immune response at the PDT treated tumor site, and to evaluate the systemic anti-tumor immune response. The long-term objective of these studies is to provide an easily administered, adjunctive, therapeutic maneuver that lacks systemic toxicity, with the potential to modulate the natural biology of colorectal cancers that have not elicited a favorable anti-tumor immune response and to improve patient survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically proven diagnosis of colorectal cancer.
2. Have clinical stage I, II, or III disease.
3. Expected survival must be greater than twelve (12) months.
4. A Karnofsky Performance Status (KPS) must be 70 or greater (Appendix I).
5. Patients must be >21 years of age.
6. No prior therapy.
7. Female patients must not be lactating and must be surgically sterile (via hysterectomy or bilateral tubal ligation), postmenopausal, or using acceptable methods of contraception if they are of child bearing potential. Female patients of childbearing potential must also have a negative serum pregnancy test.
8. Patients must be able to understand and sign an informed consent form, which must comply with U.S. regulations (U.S. 21 CFR 50) and ICH guidelines.
9. Eligible patients must have adequate initial hematologic and coagulation parameters, hemoglobin ≥ 11g/dl, platelet count >50,000, Protime and Prothrombin Time ≤ 1.5 x normal.
10. Eligible patients must have adequate bone marrow, liver and renal function: ANC > 1500/μL, Platelets >100,000 x μL, total bilirubin < the upper limit of normal (ULN), and creatinine clearance (CrCl) > 45 mL/min

Exclusion Criteria:

1. Any co-morbidity that precludes primary surgical resection of the colorectal tumor.
2. Any significant general organ system compromise including:

   * Liver function, transaminases ≥ 2 x,
   * Renal function, Cr ≥ 1.5 x upper limit of normal
   * Pulmonary function, room air O2 saturation <90%
   * Cardiovascular function, Patients with significant (Class III or IV) cardiovascular disease according to the New York Heart Association's functional criteria (Appendix II)
   * Gastrointestinal function, i.e. active inflammatory bowel disease or active peptic ulcer disease.
3. Any contraindication to repeat colonoscopy, such as idiosyncratic reactivity to conscious sedation medications.
4. Prior treatment for the diagnosis of colorectal cancer, including surgical resection.
5. Stage IV colorectal cancer, i.e. the clinical presence of metastases
6. Prior malignant diagnosis except for the basal cell epithelioma of the skin.
7. Persistent fever greater than 38 C.
8. Mineral overload syndromes for Lead, Zinc, Copper or Iron.
9. Use of any agent that modulates 5-ALA metabolism and porphyrin synthesis, e.g. St. John's Wort.
10. Required use of corticosteroids or immune suppression for any reason including an organ allograft or HIV infection
11. Patients with any acute or chronic illness including cardiovascular disease (e.g. history of atrial fibrillation or ventricular arrhythmias) or history of myocardial infarction, autoimmune state, or any psychiatric illness that in the opinion of the Investigators would compromise treatment.
12. Use of investigational drugs within 30 days of execution of the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Efficacy | 6 months
  Define biologic efficacy of PDT in relation to generation of an immune response at the tumor site and systemically. This will be measured by degree of dendritic cell infiltration into tumor and regional lymph nodes, and degree of systemic immunity directed against colon cancer antigens immediately post procedure and after 6 months.
Safety | 6 months
  Safety will be evaluated from enrollment through 6 months. This will be measured by proportion of patients completing planned surgery, proportion of patients experiencing grade 3 or 4 toxicities, and lack of observation of serious adverse events related to the study procedure.

SECONDARY OUTCOMES:
Quality of Life | 6 months after completion of participation
  Quality of life will be evaluated 6 months following completion of participation in the study
Sustained immunity | 1.5-6 months post completion of participation
  Immunologic parameters will be monitored following completion of the study as a measure of sustained immunity

CONTACTS AND LOCATIONS:
Overall Officials: Randall F Holcombe, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Edward L Nelson, MD, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - University of California, Irvine, Orange, California
  - Mounst Sinai School of Medicine, New York, New York